CLINICAL TRIAL: NCT01075282
Title: A Randomized, Open-Label, Parallel-Arm, Noninferiority Comparison of the Effects of Two Doses of LY2189265 and Insulin Glargine on Glycemic Control in Patients With Type 2 Diabetes on Stable Doses of Metformin and Glimepiride
Brief Title: A Study in Participants With Type 2 Diabetes Mellitus (AWARD-2)
Acronym: AWARD-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11374; H9X-MC-GBDB (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; dulaglutide; Metformin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY2189265 1.5 mg (Experimental): LY2189265 (Dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), once weekly for 78 weeks
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 78 weeks
  Glimepiride: at least 4 mg/day, oral, for 78 weeks
  Interventions: Drug: LY2189265; Drug: Metformin; Drug: Glimepiride
- LY2189265 0.75 mg (Experimental): LY2189265 (Dulaglutide): 0.75 milligrams (mg), subcutaneous (SC), once weekly for 78 weeks
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 78 weeks
  Glimepiride: at least 4 mg/day, oral, for 78 weeks
  Interventions: Drug: LY2189265; Drug: Metformin; Drug: Glimepiride
- Insulin Glargine (Active Comparator): Insulin Glargine: dose titration based on blood glucose measures, subcutaneous (SC), once daily for 78 weeks
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 78 weeks
  Glimepiride: at least 4 mg/day, oral, for 78 weeks
  Interventions: Drug: Insulin Glargine; Drug: Metformin; Drug: Glimepiride

INTERVENTIONS:
Drug: Insulin Glargine
  Arms: Insulin Glargine
Drug: LY2189265
  Other Names: Dulaglutide
  Arms: LY2189265 0.75 mg; LY2189265 1.5 mg
Drug: Metformin
Drug: Glimepiride

SUMMARY:
The purpose of this study is to determine if LY2189265 is effective in reducing hemoglobin A1c (HbA1c) and safe, as compared to Insulin Glargine in participants with Type 2 Diabetes. Participants must also be taking metformin and glimepiride.

DETAILED DESCRIPTION:
Rescue therapy refers to 1 of 2 types of additional therapy, each given for a different reason: any additional therapeutic intervention in participants who developed persistent, severe hyperglycemia despite full compliance with the assigned therapeutic regimen, or initiation of an alternative antihyperglycemic medication following study drug discontinuation. Participants who received rescue therapy were included in the analysis population, but only measurements obtained prior to the beginning of rescue therapy were included in specified efficacy analyses.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes not well controlled on 1, 2, or 3 oral antidiabetic medications (at least one of them must be metformin and/or a sulfonylurea)

  1. Glycosylated hemoglobin (HbA1c) greater than or equal to 7 and less than or equal to 11 if taking 1 oral antidiabetic medication
  2. HbA1c greater than or equal to 7 and less than or equal to 10 if on 2 or 3 oral antidiabetic medications
* Accept treatment with metformin and glimepiride throughout the study, as per protocol
* Willing to inject subcutaneous medication once weekly for LY2189265 or once daily for Insulin Glargine.
* Stable weight for 3 months prior to screening
* Body mass index (BMI) between 23 and 45 kilograms per square meter (kg/m^2)
* Females of child bearing potential must test negative for pregnancy at screening by serum pregnancy test and be willing to use a reliable method of birth control during the study and for 1 month following the last dose of study drug

Exclusion Criteria:

* Type 1 Diabetes
* HbA1c equal to or less than 6.5 at randomization
* Chronic insulin use
* Taking drugs to promote weight loss by prescription or over the counter
* Taking systemic steroids for greater than 14 days except for topical, eye, nasal, or inhaled
* History of Heart Failure New York Heart Classification III or IV, or acute myocardial infarction, or stroke within 2 months of screening
* Gastrointestinal (GI) problems such as diabetic gastroparesis or bariatric surgery (stomach stapling) or chronically taking drugs that directly affect GI motility
* Hepatitis or liver disease or ALT (alanine transaminase) greater than 3.0 of upper normal limit
* Acute or chronic pancreatitis of any form
* Renal disease (kidney) with a serum creatinine of greater than or equal to 1.5 milligrams per deciliter (mg/dL) for males and greater than or equal to 1.4 mg/dL for females, or a creatinine clearance of less than 60 milliliters per minute (ml/min)
* History (includes family) of type 2A or 2B Multiple Endocrine Neoplasia (MEN 2A or 2B) or medullary c-cell hyperplasia or thyroid cancer
* A serum calcitonin greater than or equal to 20 picograms per milliliter (pcg/ml) at screening
* Significant active autoimmune disease such as Lupus or Rheumatoid Arthritis
* History of or active malignancy except skin or in situ cervical or prostate cancer for within last 5 years
* Sickle cell, hemolytic anemia, or other hematological condition that may interfere with HbA1c testing
* Organ transplant except cornea
* Have enrolled in another clinical trial within the last 30 days
* Have previously signed an informed consent or participated in a LY2189265 study
* Have taken a glucagon-like peptide 1 (GLP-1) receptor agonist within the 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 2010-02; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (78):
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mendoza
- Australia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wollongong, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brisbane, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keswick, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Ringwood, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg, Victoria
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gribomont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Joinville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coquitlam, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. John's, Newfoundland and Labrador
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Markham, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mississauga, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- Croatia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Slavonski Brod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- Czechia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holešov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corbeil-Essonnes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pessac
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tours
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Greece
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Makó
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mosonmagyaróvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Székesfehérvár
- India (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aligarh
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chennai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Patna
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coatzacoalcos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuernavaca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydogoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galati
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Košice, Slovakia
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucheon-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ilsan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pusan
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ávila
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Requena
- Sweden (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsingborg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
- Taiwan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiayi City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yung-Kang, Tainan

REFERENCES:
- [Derived] Boustani MA, Pittman I 4th, Yu M, Thieu VT, Varnado OJ, Juneja R. Similar efficacy and safety of once-weekly dulaglutide in patients with type 2 diabetes aged >/=65 and <65 years. Diabetes Obes Metab. 2016 Aug;18(8):820-8. doi: 10.1111/dom.12687. Epub 2016 Jun 7. PMID 27161178
- [Derived] Yu M, Van Brunt K, Varnado OJ, Boye KS. Patient-reported outcome results in patients with type 2 diabetes treated with once-weekly dulaglutide: data from the AWARD phase III clinical trial programme. Diabetes Obes Metab. 2016 Apr;18(4):419-24. doi: 10.1111/dom.12624. Epub 2016 Feb 4. PMID 26691396
- [Derived] Giorgino F, Benroubi M, Sun JH, Zimmermann AG, Pechtner V. Efficacy and Safety of Once-Weekly Dulaglutide Versus Insulin Glargine in Patients With Type 2 Diabetes on Metformin and Glimepiride (AWARD-2). Diabetes Care. 2015 Dec;38(12):2241-9. doi: 10.2337/dc14-1625. Epub 2015 Jun 18. PMID 26089386

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2189265 1.5 mg: LY2189265 (Dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), once weekly for 78 weeks
  Metformin: at least 1500 milligram per day (mg/day), oral, for 78 weeks
  Glimepiride: at least 4 mg/day, oral, for 78 weeks
- LY2189265 0.75 mg: LY2189265 (Dulaglutide): 0.75 milligrams (mg), subcutaneous (SC), once weekly for 78 weeks
  Metformin: at least 1500 milligram per day (mg/day), oral, for 78 weeks
  Glimepiride: at least 4 mg/day, oral, for 78 weeks
- Insulin Glargine: Insulin Glargine: dose titration based on blood glucose measures, subcutaneous (SC), once daily for 78 weeks
  Metformin: at least 1500 milligram per day (mg/day), oral, for 78 weeks
  Glimepiride: at least 4 mg/day, oral, for 78 weeks
Period: Overall Study
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Started | 273 | 272 | 265 (Of 265 participants randomized to Insulin Glargine, 3 chose not to take study drug.)
Received at Least One Dose of Study Drug | 273 | 272 | 262
Completed | 242 | 243 | 238
Not Completed | 31 | 29 | 27
Not completed — Withdrawal by Subject | 11 | 7 | 11
Not completed — Adverse Event | 9 | 8 | 5
Not completed — Entry Criteria Not Met | 3 | 2 | 0
Not completed — Lost to Follow-up | 3 | 3 | 3
Not completed — Physician Decision | 3 | 3 | 3
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Treatment Non-compliance | 1 | 2 | 2
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Death | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and received at least 1 dose of LY2189265 or Insulin Glargine.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine | Total
Number analyzed (Participants) | 273 | 272 | 262 | 807
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.24 (9.76) | 56.56 (9.27) | 57.21 (9.38) | 56.66 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 136 | 128 | 393
  Male | 144 | 136 | 134 | 414
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 98 | 96 | 97 | 291
  Not Hispanic or Latino | 175 | 176 | 165 | 516
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 29 | 31 | 29 | 89
  Asian | 48 | 46 | 43 | 137
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 193 | 193 | 184 | 570
  More than one race | 2 | 1 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 13 | 13 | 12 | 38
  Slovakia | 1 | 1 | 0 | 2
  Greece | 6 | 6 | 7 | 19
  Spain | 10 | 12 | 13 | 35
  Italy | 2 | 3 | 1 | 6
  India | 30 | 27 | 27 | 84
  France | 2 | 3 | 1 | 6
  Czech Republic | 12 | 14 | 13 | 39
  Hungary | 16 | 16 | 15 | 47
  Mexico | 29 | 28 | 27 | 84
  Canada | 26 | 25 | 24 | 75
  Argentina | 55 | 54 | 54 | 163
  Belgium | 7 | 5 | 3 | 15
  Brazil | 6 | 5 | 7 | 18
  Poland | 16 | 18 | 17 | 51
  Croatia | 3 | 4 | 4 | 11
  Romania | 23 | 22 | 22 | 67
  Australia | 13 | 13 | 13 | 39
  Sweden | 2 | 0 | 1 | 3
  Korea, Republic of | 1 | 3 | 1 | 5
Body Weight [Mean (Standard Deviation); unit: kilograms] | 85.13 (17.90) | 86.18 (18.15) | 87.66 (19.62) | 86.31 (18.56)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 31.23 (5.21) | 31.51 (5.41) | 31.91 (5.76) | 31.55 (5.46)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 8.18 (1.03) | 8.13 (0.98) | 8.10 (0.95) | 8.14 (0.99)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 9.13 (6.22) | 9.28 (5.93) | 8.87 (5.98) | 9.10 (6.04)
Fasting Serum Glucose [Mean (Standard Deviation); unit: millimoles per liter (mmol/L)] | 9.16 (2.73) | 8.96 (2.70) | 9.08 (2.66) | 9.07 (2.69)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 52 Weeks Endpoint in Glycosylated Hemoglobin (HbA1c)
Description: Least Squares (LS) means were calculated using analysis of covariance (ANCOVA) with country and treatment as fixed effects and baseline HbA1c as a covariate.
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable HbA1c data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 263 | 267 | 259
percentage of glycosylated hemoglobin | -1.08 (0.06) | -0.76 (0.06) | -0.63 (0.06)
Statistical Analysis 1: Comparison: LY2189265 1.5 mg vs Insulin Glargine; The study was designed with 90% power to detect non-inferiority of LY2189265 1.5 mg vs insulin glargine on HbA1c change from baseline at the 52-week primary endpoint with a margin of 0.4%, a standard deviation of 1.3%, and a 1-sided alpha of 0.025 assuming no true difference between treatments. This corresponds to 223 participants per arm, with an assumed drop-out rate of 20%; Test type: Non-Inferiority or Equivalence — Family-wise Type I error rate was controlled by applying gatekeeping strategy; p < 0.001, ANCOVA — P-value is adjusted for multiplicity, based on tree-gatekeeping strategy. To determine significance, p-value is compared to the family-wise 1-sided Type I error of 0.025. The confidence interval is not adjusted for multiplicity; LS Mean Difference = -0.45, 95% CI 2-sided [-0.60 to -0.29]
Statistical Analysis 2: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Non-inferiority analysis; Test type: Non-Inferiority or Equivalence — Family-wise Type I error rate was controlled by applying gatekeeping strategy; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.13, 95% CI 2-sided [-0.29 to 0.02]
Statistical Analysis 3: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.45, 95% CI 2-sided [-0.60 to -0.29]
Statistical Analysis 4: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Superiority analysis; Test type: Superiority or Other; p = 0.05, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.13, 95% CI 2-sided [-0.29 to 0.02]

2. Secondary Outcome: Change From Baseline to 26 Weeks and 78 Weeks Endpoint in Glycosylated Hemoglobin (HbA1c)
Description: as for outcome 1
Time Frame: Baseline, 26 weeks, and 78 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
percent
  26 weeks (n=263, 266, 258) | -1.16 (0.06) | -0.89 (0.05) | -0.65 (0.06)
  78 weeks (n=263, 267, 259) | -0.90 (0.07) | -0.62 (0.07) | -0.59 (0.07)
Statistical Analysis 1: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Non-inferiority analysis; Test type: Non-Inferiority or Equivalence — Family-wise Type I error rate was controlled by applying gatekeeping strategy; p < 0.001, ANCOVA — Treatment comparison at 26 weeks. P-value is adjusted for multiplicity, based on tree-gatekeeping strategy, and compared to the family-wise 1-sided Type I error of 0.025. The confidence interval is not adjusted for multiplicity; LS Mean Difference = -0.51, 95% CI 2-sided [-0.65 to -0.37]
Statistical Analysis 2: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Non-inferiority analysis; Test type: Non-Inferiority or Equivalence — Family-wise Type I error rate was controlled by applying gatekeeping strategy; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.24, 95% CI 2-sided [-0.38 to -0.10]
Statistical Analysis 3: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.51, 95% CI 2-sided [-0.65 to -0.37]
Statistical Analysis 4: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.24, 95% CI 2-sided [-0.38 to -0.10]
Statistical Analysis 5: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Non-inferiority analysis; Test type: Non-Inferiority or Equivalence — Family-wise Type I error rate was controlled by applying gatekeeping strategy; p < 0.001, ANCOVA — Treatment comparison at 78 weeks. P-value is adjusted for multiplicity, based on tree-gatekeeping strategy, and compared to the family-wise 1-sided Type I error of 0.025. The confidence interval is not adjusted for multiplicity; LS Mean Difference = -0.31, 95% CI 2-sided [-0.50 to -0.13]
Statistical Analysis 6: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Non-inferiority analysis; Test type: Non-Inferiority or Equivalence — Family-wise Type I error rate was controlled by applying gatekeeping strategy; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 5]; LS Mean Difference = -0.03, 95% CI 2-sided [-0.21 to 0.15]
Statistical Analysis 7: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 5]; LS Mean Difference = -0.31, 95% CI 2-sided [-0.50 to -0.13]
Statistical Analysis 8: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Superiority analysis; Test type: Superiority or Other; p = 0.378, ANCOVA — [p-value comment as in outcome 2, analysis 5]; LS Mean Difference = -0.03, 95% CI 2-sided [-0.21 to 0.15]

3. Secondary Outcome: Number of Participants Achieving Glycosylated Hemoglobin (HbA1c) Less Than 7% at 26, 52 and 78 Weeks
Description: Number of participants achieving HbA1c levels less than 7.0% was analyzed with a logistic regression model with baseline, country, and treatment as factors included in the model.
Time Frame: 26, 52, and 78 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
participants
  26 weeks (n=263, 266, 258) | 153 | 122 | 84
  52 weeks (n=263, 267, 259) | 140 | 99 | 80
  78 weeks (n=263, 267, 259) | 129 | 91 | 79
Statistical Analysis 1: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison at 26 weeks; Odds Ratio (OR) = 4.61, 95% CI 2-sided [2.98 to 7.11]
Statistical Analysis 2: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison at 26 weeks; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.41 to 3.24]
Statistical Analysis 3: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison at 52 weeks; Odds Ratio (OR) = 3.76, 95% CI 2-sided [2.45 to 5.75]
Statistical Analysis 4: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Test type: Superiority or Other; p = 0.098, Regression, Logistic — Treatment comparison at 52 weeks; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.94 to 2.15]
Statistical Analysis 5: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison at 78 weeks; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.85 to 4.14]
Statistical Analysis 6: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Test type: Superiority or Other; p = 0.334, Regression, Logistic — Treatment comparison at 78 weeks; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.82 to 1.82]

4. Secondary Outcome: Number of Participants Achieving Glycosylated Hemoglobin (HbA1c) Less Than or Equal to 6.5% at 26, 52 and 78 Weeks
Description: Number of participants achieving HbA1c levels less than or equal to 6.5% was analyzed with a logistic regression model with baseline, country, and treatment as factors included in the model.
Time Frame: 26, 52, and 78 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
participants
  26 weeks (n=263, 266, 258) | 97 | 74 | 40
  52 weeks (n=263, 267, 259) | 71 | 60 | 35
  78 weeks (n=263, 267, 259) | 74 | 59 | 43
Statistical Analysis 1: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison at 26 weeks; Odds Ratio (OR) = 4.70, 95% CI 2-sided [2.90 to 7.63]
Statistical Analysis 2: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison at 26 weeks; Odds Ratio (OR) = 2.54, 95% CI 2-sided [1.57 to 4.11]
Statistical Analysis 3: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison at 52 weeks; Odds Ratio (OR) = 2.97, 95% CI 2-sided [1.81 to 4.85]
Statistical Analysis 4: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Test type: Superiority or Other; p = 0.004, Regression, Logistic — Treatment comparison at 52 weeks; Odds Ratio (OR) = 2.07, 95% CI 2-sided [1.26 to 3.39]
Statistical Analysis 5: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison at 78 weeks; Treatment comparison at 78 weeks; Odds Ratio (OR) = 2.27, 95% CI 2-sided [1.44 to 3.57]
Statistical Analysis 6: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Test type: Superiority or Other; p = 0.073, Regression, Logistic — Treatment comparison at 78 weeks; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.96 to 2.42]

5. Secondary Outcome: Change From Baseline to 26, 52 and 78 Weeks for Daily Mean Blood Glucose Values From the 8-point Self-monitored Blood Glucose (SMBG) Profiles
Description: The self-monitored blood glucose (SMBG) data were collected at the following 8 time points: pre-morning meal; 2 hours post-morning meal; pre-midday meal; 2 hours post-midday meal; pre-evening meal; 2 hours post-evening meal; bedtime; and 3 AM or 5 hours after bedtime. Least Squares (LS) means of the mean of the 8 time points (Daily Mean) were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable SMBG data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 231 | 242 | 228
millimoles per liter (mmol/L)
  26 weeks (n=199, 204, 190) | -1.79 (0.10) | -1.46 (0.10) | -1.58 (0.10)
  52 weeks (n=180, 185, 176) | -1.69 (0.11) | -1.32 (0.11) | -1.44 (0.11)
  78 weeks (n=172, 164, 168) | -1.55 (0.13) | -1.15 (0.12) | -1.47 (0.13)
Statistical Analysis 1: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Test type: Superiority or Other; p = 0.109, Mixed Models Analysis — Treatment comparison at 26 weeks
Statistical Analysis 2: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Test type: Superiority or Other; p = 0.335, Mixed Models Analysis — Treatment comparison at 26 weeks
Statistical Analysis 3: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Test type: Superiority or Other; p = 0.091, Mixed Models Analysis — Treatment comparison at 52 weeks
Statistical Analysis 4: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Test type: Superiority or Other; p = 0.400, Mixed Models Analysis — Treatment comparison at 52 weeks
Statistical Analysis 5: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Test type: Superiority or Other; p = 0.641, Mixed Models Analysis — Treatment comparison at 78 weeks
Statistical Analysis 6: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Test type: Superiority or Other; p = 0.055, Mixed Models Analysis — Treatment comparison at 78 weeks

6. Secondary Outcome: Change From Baseline to 52 and 78 Weeks in Updated Homeostasis Model Assessment of Beta-cell Function (HOMA2-%B) and Updated Homeostasis Model Assessment of Insulin Sensitivity (HOMA2-%S)
Description: The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance and beta (β)-cell function. HOMA2-B is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady state beta cell function (%B) as a percentage of a normal reference population (normal young adults). HOMA2-S is a computer model that uses fasting plasma insulin and glucose concentrations to estimate insulin sensitivity (%S), as percentages of a normal reference population (normal young adults). The normal reference population for both HOMA2-B and HOMA-2S were set at 100%. Least Squares (LS) means of change from baseline of C-peptide based HOMA2-%B and HOMA2-%S were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 with evaluable HOMA2-%B or HOMA2-%S data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg
Number analyzed (Participants) | 222 | 230
percentage of HOMA2
  HOMA2-%B, 52 weeks (n=175, 181) | 29.95 (4.61) | 24.60 (4.51)
  HOMA2-%B, 78 weeks (n=167, 165) | 28.54 (4.78) | 15.66 (4.75)
  HOMA2-%S, 52 weeks (n=175,181) | -2.89 (1.21) | -2.66 (1.19)
  HOMA2-%S, 78 weeks (n=167, 165) | -2.64 (1.23) | -3.62 (1.23)

7. Secondary Outcome: Change From Baseline to 52 and 78 Weeks in Glucagon Concentration
Description: Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country and treatment as fixed effects and baseline as a covariate.
Time Frame: Baseline, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable glucagon data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: picomoles per liter (pmol/L)
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 235 | 235 | 232
picomoles per liter (pmol/L)
  52 weeks (n=232, 231, 228) | -3.91 (0.47) | -3.31 (0.47) | -3.85 (0.47)
  78 weeks (n=235, 235, 232) | -3.57 (0.47) | -3.37 (0.47) | -3.65 (0.47)

8. Secondary Outcome: Change From Baseline to 26, 52 and 78 Weeks for Body Weight
Description: as for outcome 7
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable body weight data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 272 | 270 | 259
kilogram (kg)
  26 weeks | -1.82 (0.20) | -1.47 (0.20) | 1.01 (0.20)
  52 weeks | -1.87 (0.24) | -1.33 (0.24) | 1.44 (0.24)
  78 weeks | -1.96 (0.26) | -1.54 (0.26) | 1.28 (0.26)
Statistical Analysis 1: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 26 weeks; LS Mean Difference = 2.83, 95% CI 2-sided [2.33 to 3.33]
Statistical Analysis 2: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 26 weeks; LS Mean Difference = 2.48, 95% CI 2-sided [1.99 to 2.99]
Statistical Analysis 3: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 52 weeks; LS Mean Difference = 3.31, 95% CI 2-sided [2.71 to 3.90]
Statistical Analysis 4: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 52 weeks; LS Mean Difference = 2.77, 95% CI 2-sided [2.17 to 3.36]
Statistical Analysis 5: Comparison: LY2189265 1.5 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 78 weeks; LS Mean Difference = 3.24, 95% CI 2-sided [2.59 to 3.89]
Statistical Analysis 6: Comparison: LY2189265 0.75 mg vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 78 weeks; LS Mean Difference = 2.82, 95% CI 2-sided [2.17 to 3.46]

9. Secondary Outcome: Change From Baseline to 26, 52 and 78 Weeks for Body Mass Index
Description: Body mass index (BMI) is an estimate of body fat based on body weight divided by height squared. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable BMI data.
Measure: Least Squares Mean (Standard Error); unit: kilograms per square meter (kg/m^2)
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
kilograms per square meter (kg/m^2)
  26 weeks (n=257, 261, 245) | -0.64 (0.07) | -0.50 (0.07) | 0.44 (0.07)
  52 weeks (n=250, 252, 238) | -0.64 (0.08) | -0.39 (0.08) | 0.62 (0.08)
  78 weeks (n=246, 244, 238) | -0.64 (0.09) | -0.39 (0.09) | 0.59 (0.10)

10. Secondary Outcome: Change From Baseline to 26, 52 and 78 Weeks in the EuroQol 5 Dimension
Description: The European Quality of Life - 5 dimensions (EQ-5D) questionnaire is a generic, multidimensional, health-related, quality-of-life instrument. It consists of 2 parts: the first part assesses 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that have 3 possible levels of response (no problem, some problem, or extreme problem). These dimensions are converted into a weighted health-state Index Score. The EQ-5D United Kingdom (UK) score ranges from -0.59 to 1.0, where a score of 1.0 indicates perfect health and negative values are valued as worse than dead. The second part of the questionnaire consists of a 100-mm visual analog scale (VAS) on which the participants rated their perceived health state on that day from 0 (worst imaginable health state) to 100 (best imaginable health). Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) and adjusted by treatment, country, and baseline.
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable EQ-5D data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
units on a scale
  EQ-5D UK, 26 weeks (n=257, 254, 249) | 0.01 (0.01) | 0.00 (0.01) | -0.01 (0.01)
  EQ-5D UK, 52 weeks (n=259, 260, 253) | 0.01 (0.01) | 0.00 (0.01) | -0.04 (0.01)
  EQ-5D UK, 78 weeks (n=259, 260, 253) | 0.01 (0.01) | 0.00 (0.01) | 0.00 (0.01)
  VAS, 26 weeks (n=253, 252, 243) | 3.3 (0.83) | 3.4 (0.84) | 0.8 (0.86)
  VAS, 52 weeks (n=260, 258, 252) | 3.2 (0.85) | 2.3 (0.85) | 1.1 (0.88)
  VAS, 78 weeks (n=260, 258, 252) | 3.8 (0.85) | 3.2 (0.85) | 2.2 (0.89)

11. Secondary Outcome: Change From Baseline to 26, 52 and 78 Weeks in the Impact of Weight on Activities of Daily Living
Description: The Impact of Weight on Activities of Daily Living questionnaire (renamed the Ability to Perform Physical Activities of Daily Living Questionnaire [APPADL]) contains 7 items that assess how difficult it is for participants to engage in certain activities considered to be integral to normal daily life, such as walking, standing and climbing stairs. Items are scored on a 5-point numeric rating scale where 5 = "not at all difficult" and 1 = "unable to do". The individual scores from all 7 items are summed and a single total score is calculated and may range between 7 and 35. A higher score indicates better ability to perform activities of daily living. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country and treatment as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable APPADL data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 260
units on a scale
  26 weeks (n=256, 256, 248) | 0.7 (0.30) | 0.1 (0.30) | -0.3 (0.30)
  52 weeks (n=260, 261, 249) | 0.9 (0.31) | 0.4 (0.31) | -0.6 (0.32)
  78 weeks (n=260, 261, 249) | 1.0 (0.31) | 0.3 (0.31) | -0.3 (0.32)

12. Secondary Outcome: Change From Baseline to 26, 52 and 78 Weeks in the Impact of Weight on Self-Perception
Description: The Impact of Weight on Self-Perception (IW-SP) questionnaire contains 3 items that assess how often the participants' body weight affects how happy they are with their appearance and how often they feel self-conscious when out in public. Items are scored on a 5-point numeric rating scale where 5 = never and 1 = always. A single total score is calculated by summing the scores for all 3 items. Total score ranges between 3 and 15, where a higher score is indicative of better self-perception. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country and treatment as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable IW-SP data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
units on a scale
  26 weeks (n=258, 258, 251) | 0.1 (0.16) | 0.2 (0.16) | -0.1 (0.16)
  52 weeks (n=260, 261, 252) | 0.5 (0.16) | 0.2 (0.16) | 0.1 (0.16)
  78 weeks (n=260, 261, 252) | 0.5 (0.16) | 0.3 (0.15) | 0.1 (0.16)

13. Secondary Outcome: Change From Baseline to 26, 52 and 78 Weeks in the Low Blood Sugar Survey
Description: The Low Blood Sugar Survey (LBSS) contains 33 items comprised of 2 subscales (behavior and worry), each of which is rated on a 5-point numeric rating scale from 0 (never) to 4 (almost always). It captures behavioral changes associated with the concerns and experiences of hypoglycemia and the degree to which participants are worried about certain aspects associated with hypoglycemia during the previous 4 weeks. The behavior (or avoidance) subscale has 15 items, and the worry (or affect) subscale has 18 items. Subscale scores are calculated by summing participant responses to items (behavior range 0-60; worry range 0-72). A total score is calculated as the sum of both subscales (range 0-132). Higher scores indicate greater negative impact on subscales and total score. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country and treatment as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable LBSS data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 270 | 271 | 255
units on a scale
  26 weeks (n=255, 255, 244) | -2.8 (0.95) | -2.4 (0.96) | 0.3 (0.98)
  52 weeks (n=258, 259, 245) | -4.2 (0.83) | -4.1 (0.83) | -1.0 (0.86)
  78 weeks (n=258, 259, 245) | -4.6 (0.82) | -4.7 (0.82) | -2.0 (0.85)

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events at 26, 52 and 78 Weeks
Description: A treatment-emergent adverse event (TEAE) was defined as an event that first occurs or worsens (increases in severity) after baseline regardless of causality or severity. The number of participants with one or more TEAE is summarized cumulatively at 26, 52, and 78 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine. The number of participants with at least 1 TEAE is reported.
Measure: Number; unit: participants
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
participants
  26 weeks | 160 | 146 | 137
  52 weeks | 189 | 175 | 175
  78 weeks | 201 | 188 | 192

15. Secondary Outcome: Number of Self-reported Hypoglycemic Events at 26, 52 and 78 Weeks
Description: Hypoglycemic events (HE) were classified as severe (defined as episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a plasma glucose level of =<3.9 mmol/L), asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of =<3.9 mmol/L), nocturnal (defined as any hypoglycemic event that occurred between bedtime and waking), or probable symptomatic (defined as events during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination). The number of self-reported hypoglycemic events is summarized cumulatively at 26, 52, and 78 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine.
Measure: Number; unit: events
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
events
  Severe HE, 26 weeks | 1 | 0 | 1
  Severe HE, 52 weeks | 1 | 0 | 2
  Severe HE, 78 weeks | 2 | 0 | 2
  Documented symptomatic HE, 26 weeks | 311 | 315 | 447
  Documented symptomatic HE, 52 weeks | 515 | 444 | 789
  Documented symptomatic HE, 78 weeks | 607 | 515 | 1033
  Asymptomatic HE, 26 weeks | 500 | 484 | 609
  Asymptomatic HE, 52 weeks | 757 | 709 | 1093
  Asymptomatic HE, 78 weeks | 884 | 911 | 1358
  Nocturnal HE, 26 weeks | 145 | 117 | 240
  Nocturnal HE, 52 weeks | 185 | 147 | 519
  Nocturnal HE, 78 weeks | 215 | 184 | 635
  Probable symptomatic HE, 26 weeks | 11 | 19 | 20
  Probable symptomatic HE, 52 weeks | 17 | 24 | 22
  Probable symptomatic HE, 78 weeks | 20 | 28 | 26

16. Secondary Outcome: Rate of Self-reported Hypoglycemic Events at 26, 52 and 78 Weeks
Description: Hypoglycemic events (HE) were classified as severe (defined as episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a plasma glucose level of =<3.9 mmol/L), asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of =<3.9 mmol/L), nocturnal (defined as any hypoglycemic event that occurred between bedtime and waking), or probable symptomatic (defined as events during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination). The 1-year adjusted rate of hypoglycemic events is summarized cumulatively at 26, 52, and 78 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine.
Measure: Mean (Standard Deviation); unit: events per participant per year
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
events per participant per year
  Severe HE, 26 weeks | 0.01 (0.12) | 0.00 (0.00) | 0.01 (0.12)
  Severe HE, 52 weeks | 0.00 (0.06) | 0.00 (0.00) | 0.01 (0.09)
  Severe HE, 78 weeks | 0.01 (0.06) | 0.00 (0.00) | 0.01 (0.06)
  Documented symptomatic HE, 26 weeks | 2.35 (5.41) | 2.52 (6.42) | 3.64 (6.63)
  Documented symptomatic HE, 52 weeks | 2.03 (4.16) | 1.97 (5.31) | 3.34 (5.91)
  Documented symptomatic HE, 78 weeks | 1.67 (3.58) | 1.66 (4.96) | 3.03 (5.63)
  Asymptomatic HE, 26 weeks | 3.79 (8.01) | 3.58 (7.70) | 4.82 (11.43)
  Asymptomatic HE, 52 weeks | 3.08 (6.97) | 2.68 (5.40) | 4.41 (8.72)
  Asymptomatic HE, 78 weeks | 2.56 (5.90) | 2.38 (4.95) | 3.80 (7.24)
  Nocturnal HE, 26 weeks | 1.23 (3.84) | 0.96 (3.53) | 1.86 (4.84)
  Nocturnal HE, 52 weeks | 0.90 (3.13) | 0.65 (2.65) | 2.07 (4.67)
  Nocturnal HE, 78 weeks | 0.77 (2.97) | 0.59 (2.47) | 1.81 (4.12)
  Probable symptomatic HE, 26 weeks | 0.08 (0.59) | 0.14 (1.39) | 0.15 (0.87)
  Probable symptomatic HE, 52 weeks | 0.07 (0.40) | 0.09 (0.99) | 0.08 (0.47)
  Probable symptomatic HE, 78 weeks | 0.05 (0.32) | 0.07 (0.67) | 0.07 (0.37)

17. Secondary Outcome: Number of Participants Requiring Additional Intervention Due to Hyperglycemia at 26, 52 and 78 Weeks
Description: Additional intervention was defined as any additional therapeutic intervention in participants who developed persistent, severe hyperglycemia despite full compliance with the assigned therapeutic regimen, or initiation of an alternative antihyperglycemic medication following study drug discontinuation. The number of participants requiring additional intervention due to hyperglycemia is summarized cumulatively at 26, 52, and 78 weeks.
Time Frame: 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine.
Measure: Number; unit: participants
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
participants
  26 weeks | 2 | 4 | 0
  52 weeks | 11 | 20 | 8
  78 weeks | 24 | 34 | 16

18. Secondary Outcome: Change From Baseline to 26, 52 and 78 Weeks on Pancreatic Enzymes
Description: Amylase (total and pancreas-derived) and lipase concentrations were measured.
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable pancreatic enzyme data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: units/liter
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 271 | 269 | 259
units/liter
  Amylase (total), 26 weeks | 4.000 [-4.000 to 13.000] | 4.000 [-3.000 to 11.000] | 2.000 [-5.000 to 8.000]
  Amylase (total), 52 weeks | 4.000 [-4.000 to 11.000] | 5.000 [-3.000 to 13.000] | 3.000 [-5.000 to 9.000]
  Amylase (total), 78 weeks | 4.000 [-4.000 to 13.000] | 4.000 [-3.000 to 12.000] | 1.000 [-7.000 to 9.000]
  Amylase (pancreas-derived), 26 weeks | 3.000 [-1.000 to 8.000] | 3.000 [0.000 to 7.000] | 1.000 [-2.000 to 4.000]
  Amylase (pancreas-derived), 52 weeks | 3.000 [-1.000 to 8.000] | 3.000 [-1.000 to 7.000] | 1.000 [-2.000 to 6.000]
  Amylase (pancreas-derived), 78 weeks | 2.000 [-2.000 to 7.000] | 2.000 [-1.000 to 7.000] | 0.000 [-3.000 to 4.000]
  Lipase, 26 weeks | 5.000 [-4.000 to 15.000] | 5.000 [-1.000 to 15.000] | -1.000 [-6.000 to 5.000]
  Lipase, 52 weeks | 4.000 [-3.000 to 12.000] | 4.000 [-2.000 to 11.000] | -1.000 [-8.000 to 6.000]
  Lipase, 78 weeks | 4.000 [-3.000 to 14.000] | 4.000 [-1.000 to 13.000] | -2.000 [-8.000 to 5.000]

19. Secondary Outcome: Number of Participants With Adjudicated Pancreatitis at 26, 52 and 78 Weeks
Description: The number of participants with pancreatitis confirmed by adjudication is summarized cumulatively at 26, 52, and 78 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine.
Measure: Number; unit: participants
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
participants
  26 weeks | 1 | 1 | 0
  52 weeks | 2 | 1 | 0
  78 weeks | 2 | 1 | 0

20. Secondary Outcome: Change From Baseline to 26, 52 and 78 Weeks on Serum Calcitonin
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable serum calcitonin data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
picogram/milliliter
  26 weeks (n=266, 267, 258) | 0.163 (1.31) | 0.097 (1.20) | 0.149 (1.30)
  52 weeks (n=266, 269, 259) | 0.128 (1.20) | 0.132 (1.32) | 0.176 (1.62)
  78 weeks (n=267, 269, 259) | 0.086 (1.31) | 0.035 (1.20) | 0.151 (1.73)

21. Secondary Outcome: Number of Participants With Adjudicated Cardiovascular Events at 26, 52 and 78 Weeks
Description: Information on cardiovascular (CV) risk factors was collected at baseline. Data on any new CV event was prospectively collected using a CV event electronic case report form. At prespecified visits, participants were asked about any new CV event. Deaths and nonfatal cardiovascular adverse events (AEs) were adjudicated by a committee of physicians with cardiology expertise external to the Sponsor. The nonfatal cardiovascular AEs to be adjudicated include myocardial infarction, hospitalization for unstable angina, hospitalization for heart failure, coronary interventions (such as coronary artery bypass graft or percutaneous coronary intervention), and cerebrovascular events including cerebrovascular accident (stroke) and transient ischemic attack. The number of participants with adjudicated CV events is summarized cumulatively at 26, 52, and 78 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine.
Measure: Number; unit: participants
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
participants
  Any CV event, 26 weeks | 2 | 1 | 3
  Any fatal CV event, 26 weeks | 0 | 0 | 0
  Any non-fatal CV event, 26 weeks | 2 | 1 | 3
  Any CV event, 52 weeks | 3 | 4 | 6
  Any fatal CV event, 52 weeks | 0 | 0 | 1
  Any non-fatal CV event, 52 weeks | 3 | 4 | 5
  Any CV event, 78 week | 3 | 6 | 9
  Any fatal CV event, 78 week | 0 | 1 | 1
  Any non-fatal CV event, 78 week | 3 | 6 | 8

22. Secondary Outcome: Change in Baseline to 26, 52 and 78 Weeks on Pulse Rate
Description: Sitting pulse rate was measured. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable sitting pulse rate data.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
beats per minute (bpm)
  26 weeks (n=257, 260, 245) | 1.56 (0.49) | 0.74 (0.48) | -1.21 (0.50)
  52 weeks (n=250, 252, 240) | 1.29 (0.50) | 0.51 (0.49) | -0.52 (0.51)
  78 weeks (n=246, 244, 238) | 1.31 (0.50) | 0.61 (0.50) | -0.91 (0.51)

23. Secondary Outcome: Change From Baseline to 26, 52, and 78 Weeks on Blood Pressure
Description: Sitting systolic blood pressure (SBP) and sitting diastolic blood pressure (DBP) were measured. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable blood pressure data.
Measure: Least Squares Mean (Standard Error); unit: milliliter of mercury (mmHG)
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
milliliter of mercury (mmHG)
  SBP, 26 weeks (n=257, 261, 245) | -1.28 (0.78) | -1.60 (0.78) | -0.03 (0.80)
  SBP, 52 weeks (n=250, 252, 240) | 0.17 (0.81) | 0.09 (0.80) | 0.51 (0.83)
  SBP, 78 weeks (n=246, 244, 238) | -0.70 (0.85) | -0.59 (0.85) | 0.51 (0.87)
  DBP, 26 weeks (n=257, 261, 245) | -0.16 (0.49) | -0.17 (0.48) | -0.29 (0.50)
  DBP, 52 weeks (n=250, 252, 240) | -0.26 (0.48) | -0.19 (0.47) | -0.93 (0.49)
  DBP, 78 weeks (n=246, 244, 238) | -0.44 (0.52) | -0.36 (0.52) | -1.04 (0.53)

24. Secondary Outcome: Change From Baseline to 26, 52 and 78 Weeks on Electrocardiogram Parameters, Heart Rate
Description: Electrocardiogram (ECG) heart rate was measured. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable ECG heart rate data.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 270 | 271 | 260
beats per minute (bpm)
  26 weeks (n=241, 247, 231) | 2.64 (0.539) | 0.90 (0.529) | -1.24 (0.549)
  52 weeks (n=232, 242, 231) | 2.41 (0.564) | 0.38 (0.551) | -1.01 (0.568)
  78 weeks (n=223, 222, 225) | 2.49 (0.592) | 0.47 (0.588) | -0.26 (0.594)

25. Secondary Outcome: Change From Baseline to 26, 52 and 78 Weeks on Electrocardiogram Parameters, Fridericia Corrected QT (QTcF) Interval and PR Interval
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTc = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between two R waves. PR is the interval between the P wave and the QRS complex. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 78 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable ECG QTcF or PR Interval data.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Number analyzed (Participants) | 273 | 272 | 262
milliseconds (msec)
  QTcF interval, 26 weeks (n=240, 245, 229) | -1.71 (0.939) | -0.10 (0.926) | 1.24 (0.962)
  QTcF interval, 52 weeks (n=231, 240, 228) | 1.55 (1.074) | 1.34 (1.054) | 3.70 (1.088)
  QTcF interval, 78 weeks (n=221, 220, 222) | 1.66 (1.045) | 3.44 (1.039) | 4.44 (1.053)
  PR interval, 26 weeks (n=240, 245, 229) | 2.78 (0.849) | 2.33 (0.836) | 1.24 (0.873)
  PR interval, 52 weeks (n=230, 240, 227) | 2.61 (0.853) | 1.88 (0.835) | 1.50 (0.868)
  PR interval, 78 weeks (n=221, 220, 222) | 2.62 (1.034) | 3.27 (1.026) | 1.21 (1.043)

26. Secondary Outcome: Number of Participants With LY2189265 Antibodies at 26, 52, 78 Weeks and 4 Weeks After Last Dose of Study Drug (83 Weeks Maximum)
Description: LY2189265 (Dulaglutide) anti-drug antibodies (ADA) were assessed at baseline, 26, 52, and 78 weeks, and at the safety follow-up visit 30 days after study drug discontinuation (83 weeks). The number of participants with initial postbaseline detection of treatment emergent (defined as a 4-fold increase in the ADA titer from baseline) LY2189265 ADA at each time point were summarized.
Time Frame: Baseline, 26, 52, 78, and 83 weeks
Population: Participants who received at least one dose of LY2189265 with evaluable LY2189265 ADA data.
Measure: Number; unit: participants
Groups:
- LY2189265 1.5 mg and 0.75 mg: LY2189265 (Dulaglutide): 1.5 milligrams (mg) or 0.75 mg, subcutaneous (SC), once weekly for 78 weeks
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 78 weeks
  Glimepiride: at least 4 mg/day, oral, for 78 weeks
Arm/Group | LY2189265 1.5 mg and 0.75 mg
Number analyzed (Participants) | 539
participants
  26 weeks | 11
  52 weeks | 3
  78 weeks | 1
  83 weeks | 0

ADVERSE EVENTS:
Arm/Group | LY2189265 1.5 mg | LY2189265 0.75 mg | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 32/273 | 28/272 | 33/262
Other Adverse Events (participants affected / at risk) | 199/273 | 190/272 | 187/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2189265 1.5 mg (N=273) | LY2189265 0.75 mg (N=272) | Insulin Glargine (N=262)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) — One event resulted in death in 0.75 mg LY2189265 arm
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) — event resulted in death
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2)
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Hepatitis e (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0/129 (0) | 0/136 (0) | 1/128 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enzymes increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Metabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/129 (0) | 1/136 (1) | 0/128 (0)
Prostate cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/144 (1) | 0/136 (0) | 0/134 (0)
Testicular seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/144 (0) | 1/136 (1) | 0/134 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/129 (0) | 0/136 (0) | 1/128 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal cord ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — event resulted in death
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Meniscus removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Femoral arterial stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2189265 1.5 mg (N=273) | LY2189265 0.75 mg (N=272) | Insulin Glargine (N=262)
Abdominal pain (Gastrointestinal disorders) | 12 (14) | 3 (3) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 14 (17) | 9 (11) | 2 (2)
Constipation (Gastrointestinal disorders) | 12 (12) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 29 (44) | 26 (36) | 15 (20)
Dyspepsia (Gastrointestinal disorders) | 19 (20) | 9 (10) | 6 (22)
Nausea (Gastrointestinal disorders) | 42 (56) | 22 (33) | 4 (4)
Vomiting (Gastrointestinal disorders) | 18 (23) | 10 (19) | 3 (3)
Bronchitis (Infections and infestations) | 9 (10) | 7 (8) | 14 (19)
Influenza (Infections and infestations) | 12 (13) | 13 (16) | 14 (17)
Nasopharyngitis (Infections and infestations) | 16 (21) | 12 (16) | 24 (27)
Upper respiratory tract infection (Infections and infestations) | 15 (21) | 11 (18) | 17 (22)
Urinary tract infection (Infections and infestations) | 12 (19) | 17 (24) | 15 (18)
Viral infection (Infections and infestations) | 4 (4) | 4 (4) | 8 (11)
Pancreatic enzymes increased (Investigations) | 13 (28) | 9 (11) | 4 (7)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 12 (14) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 9 (9) | 8 (8) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (9) | 12 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 11 (11) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (12) | 10 (11) | 3 (3)
Dizziness (Nervous system disorders) | 9 (9) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 22 (38) | 9 (9) | 13 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 8 (8) | 6 (7)
Hypertension (Vascular disorders) | 12 (12) | 13 (13) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days